CLINICAL TRIAL: NCT06971315
Title: Impact of Vitamin C on Pain Detection and Tolerance Threshold: a Double-blind Randomized Controlled Trial
Brief Title: Impact of Vitamin C on Pain Detection and Tolerance Threshold
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Raoul Daoust, Dr Emergency Medicine, Professor, Clinician Researcher, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2025-2991
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Pain, Acute
Keywords: Vitamin C; Algometer; Pain detection; Pain threshold
MeSH Terms: conditions — Acute Pain | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Three doses of 900 mg of vitamin C taken orally every 12 hours for 24 hours (baseline, 12 hours and 24 hours)
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Three doses of 900 mg of placebo taken orally every 12 hours for 24 hours (baseline, 12 hours and 24 hours)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — Three doses of 900 mg vitamin C taken orally (baseline, 12 hours and 24 hours)
  Arms: Vitamin C
Other: Placebo — Three doses of 900 mg placebo taken orally (baseline, 12 hours and 24 hours)
  Arms: Placebo

SUMMARY:
Non-opioid treatments are increasingly sought after for managing acute pain. Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) (e.g., Advil, Motrin, Naproxen) combined with acetaminophen (e.g., Tylenol) have become an alternative for relieving acute pain. However, many patients cannot tolerate or have contraindications to NSAIDs and acetaminophen.

There is therefore an urgent need for studies evaluating the analgesic effects of vitamin C in the context of acute pain. Our study is conducted with healthy volunteer participants receiving either vitamin C or a placebo to assess the analgesic effect of vitamin C by comparing pain detection and tolerance thresholds.

DETAILED DESCRIPTION:
Opioid-free treatments are increasingly sought for acute pain and NSAIDs have become an alternative to treat acute MSK pain and are often administered in addition to acetaminophen. However, NSAIDs can produce important adverse events and are contraindicated in many patients with comorbidities (e.g., heart disease, renal failure). Similarly, acetaminophen is contraindicated in patients with active liver disease or severe hepatic impairment.

Vitamin C has shown opioid sparing and anti-inflammatory effects mostly in postoperative contexts. Vitamin C has also demonstrated very low toxicity and rare contraindications at the dosage used in this study. Demonstrating that vitamin C increases pain detection and tolerance thresholds, thereby exhibiting an analgesic effect, could offer a valuable alternative or adjunct for patients who cannot tolerate or have contraindications to NSAIDs or acetaminophen, helping to reduce opioid use. With an aging population, the number of affected patients is expected to rise significantly.

The primary outcome is the pressure pain detection threshold (PPDT) measured with an algometer one to three hours after the last dose of the study drug (24 hours after the first dose of vitamin C or placebo).

Secondary outcomes are PPDT one to three hours after the first study drug dose, PPTT one to three hours after the initial dose and last dose of the study drug, and adverse events from the algometer or the vitamin C.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 to 65 years old;
2. No acute or chronic pain;
3. No pain medication;
4. French or English-speaking

Exclusion Criteria:

1. Currently using vitamin C supplements;
2. Pain in the last week or active cancer;
3. Unavailable for follow-up;
4. Allergy to milk (lactose in the placebo), or vitamin C,
5. Treated with cyclosporine or warfarin (interaction with vitamin C);
6. Pre-existing oxalate nephropathy, liver cirrhosis or hemochromatosis;
7. Evidence of joint or overlying skin infection in the areas of testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pressure pain detection threshold (PPDT) | 24 hours
  Pressure pain detection threshold (PPDT) measured with an algometer one to three hours after the last dose of the study drug (24 hours after the first dose of vitamin C or placebo).

SECONDARY OUTCOMES:
Pressure pain detection threshold one to three hours after the first study drug dose | 1 hours
  Pressure pain detection threshold (PPDT) measured with an algometer one to three hours after the first dose of the study drug
Pressure pain tolerance threshold (PPTT) one to three hours after the last dose of the study drug | 24 hours
  Pressure pain tolerance threshold (PPTT) measured with an algometer one to three hours after the last dose of the study drug
Pressure pain tolerance threshold (PPTT) one to three hours after the first dose of the study drug | 1 hour
  Pressure pain tolerance threshold (PPTT) measured with an algometer one to three hours after the first dose of the study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada